CLINICAL TRIAL: NCT06767852
Title: the Risk Prediction Model of MACE After PCI in Patients With AMI Based on Multimodal Machine Learning and the Effect of Digital Therapeutics for Cardiac Rehabilitation
Brief Title: Risk Prediction Model of MACE in Patients With AMI Based on Multi-modal Machine Learning
Status: Not yet recruiting | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Chen Leilei, Chief Physician, The First Affiliated Hospital with Nanjing Medical University
Other Study IDs: MPAMI
Record Dates: First submitted 2024-12-30; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Acute Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A prospective, multicenter, observational study is adopted, with Jiangsu Provincial People's Hospital as the leading unit, and the other 13 Hospitals as cooperative units.

DETAILED DESCRIPTION:
The deployment of an integrated cardiac rehabilitation management platform from the hospital to the outside of the hospital is uniformly arranged, and based on this platform, a study on the construction of a MACE prediction model and disease risk stratification for patients with acute myocardial infarction after PCI is carried out. It is planned to include 655 inpatients after PCI for acute myocardial infarction. Among them, the leading unit completes the enrollment and follow-up of 44 patients, and each cooperative unit completes the enrollment and follow-up of 47 patients, and competitive enrollment is allowed.

ELIGIBILITY:
Inclusion Criteria:

* Meeting the diagnostic criteria of AMI;

  * Ages 18 - 75 years old;

    * Meeting the indications for emergency PCI surgery, with informed consent and voluntarily undergoing PCI treatment; ④ Accurate and complete clinical relevant data; ⑤ First diagnosis and treatment; ⑥ All patients were given unified antiplatelet therapy after the operation; ⑦ All patients were followed up for 12 months after the operation.

Exclusion Criteria:

* With malignant tumors, infections and other diseases;

  * Blood diseases, immune system diseases, severe liver and kidney function disorders; ③ With other heart diseases such as heart failure; ④ Patients undergoing surgical treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 - 75 years old who have undergone PCI after acute myocardial infarction.
Sampling Method: Probability Sample
Enrollment: 655 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
6-minute walk test (6MWT) | 12 months
  The test requirements refer to the guidelines formulated by the American Thoracic Society. Instruct the patient to walk back and forth on a 30-meter-long corridor at the fastest speed. Once there are obvious symptoms such as chest tightness, dizziness, and breathing difficulties, the experiment should be stopped immediately, and the walking distance of the patient within 6 minutes should be detected and recorded after the experiment.
Cardiopulmonary exercise testing (CPET) | 12 months
  Cardiopulmonary exercise testing (CPET) refers to a method of examination that, under a gradually increasing exercise load, measures a series of indicator changes in the human body, including gas metabolism, heart rate, blood pressure, blood oxygen saturation, and electrocardiogram, from the resting state to the maximum exertion state during exercise and then back to the resting state. It records the corresponding symptoms that occur in the subjects during the testing process, objectively reflecting the physiological and pathological changes and the degree of functional impairment that occur at different load levels, thereby comprehensively evaluating the overall function and reserve capacity of organ systems such as the heart and lungs. The protocol used in this study is a symptom-limited incremental exercise test using a treadmill.
electrocardiogram | At the time of enrollment
  24-hour physiological data monitoring: Wear a wearable device, and the monitoring time is from 8:00 am to 8:00 am the next day. Collect physiological signals such as electrocardiogram to evaluate heart rate variability.
breathing and blood oxygen | At the time of enrollment
  24-hour physiological data monitoring: Wear a wearable device, and the monitoring time is from 8:00 am to 8:00 am the next day. Collect physiological signals such as blood oxygen to evaluate breathing patterns, sleep breathing events and sleep stagess.
Major Adverse Cardiovascular Events (MACE) | 12 months
  Major Adverse Cardiovascular Events (MACE): Major Adverse Cardiovascular Events include heart failure, cardiovascular death, arrhythmia, atrial fibrillation, ventricular tachycardia, all-cause mortality, readmission, cardiogenic shock, target vessel revascularization, new or worsening myocardial infarction, non-fatal stroke, etc.

SECONDARY OUTCOMES:
Barthel Index | 12 months
  Barthel Index: The ability of daily living self-care is evaluated by the Barthel Index, which consists of 10 items, including eating, bathing, grooming, dressing, bowel control, bladder control, toileting, transfer from bed to chair, walking, and going up and down stairs. The total score ranges from 0 to 100. The higher the score, the better the self-care ability. A score of 100 indicates complete self-care.
Left ventricular ejection fraction, LVEF | 12 months
  The patient's cardiac function is detected by echocardiography. The patient is in the supine position, and the probe scans the parasternal long-axis view of the left ventricle, the apical four-chamber view, the two-chamber view, the short-axis view of the ventricle, etc. The left ventricular ejection fraction (LVEF)are determined. The value is obtained by calculating the average of three consecutive cardiac cycles in the apical four-chamber view using the modified Simpson's rule.
the assessment of the Generalized Anxiety Disorder 7-item scale (GAD-7) | 12 months
  Anxiety is assessed using the Generalized Anxiety Disorder 7-item scale (GAD-7). A total score of ≥5 in the assessment result is positive, indicating the possible presence of anxiety. Among them, a score of 5 - 9 may indicate mild anxiety, 10 - 14 may indicate moderate anxiety, and 15 - 21 may indicate severe anxiety.
the assessment of the Patient Health Questionnaire-9 (PHQ-9) | 12 months
  Depression is assessed using the Patient Health Questionnaire-9 (PHQ-9). A total score of ≥5 in the assessment result is positive, indicating the possible presence of depressive mood. Among them, a score of 5 - 9 may indicate mild depression, 10 - 14 may indicate moderate depression, and 15 - 27 may indicate severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: Xiangqing Kong, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- the First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China